CLINICAL TRIAL: NCT01863745
Title: An Open Label, Multi-center Nilotinib Roll-over Protocol for Patients Who Have Completed a Previous Novartis-sponsored Nilotinib Study and Are Judged by the Investigator to Benefit From Continued Nilotinib Treatment
Brief Title: Nilotinib Roll-over Protocol for Patients in Novartis-sponsored Nilotinib Study and Benefiting From Nilotinib Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107A1201
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-07

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: gastrointestinal stromal tumors; gastrointestinal,; stromal,; tumors,; GIST,; AMN107,; nilotinib
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Neoplasms | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nilotinib (Experimental): The starting dose of nilotinib was same as the last dose given in the parent nilotinib study. After this, the dose of nilotinib was based on the investigator's judgment. The total daily dose was up to 800 mg.
  Interventions: Drug: nilotinib

INTERVENTIONS:
Drug: nilotinib — Nilotinib was administered daily as hard gelatin capsules for oral use. The starting dose of nilotinib was same as the last dose given in the parent nilotinib study. After this, the dose of nilotinib was based on the investigator's judgment. The total daily dose was up to 800 mg.

SUMMARY:
The purpose of this study is to collect and assess long-term safety of nilotinib in patients who are on nilotinib treatment in a Novartis-sponsored, Oncology Clinical Development & Medical Affairs study and are benefiting from the treatment as judged by the investigator.

DETAILED DESCRIPTION:
This was an open label, multi-center, phase II study to collect and assess long-term safety of nilotinib to patients treated in Novartis sponsored clinical studies (NCT00785785 and NCT00718562) and who were benefiting from treatment with nilotinib.

There was no screening period for this study. At the enrolment visit the patient was consented to the study and eligible patients started their treatment with nilotinib.

ELIGIBILITY:
Inclusion Criteria:

* Patient is currently enrolled in a Novartis-sponsored, Clinical study receiving nilotinib and benefiting from the treatment with nilotinib, as determined by the investigator

Exclusion Criteria:

* Patient has been permanently discontinued from nilotinib treatment in the parent study due to unacceptable toxicity, non-compliance to study procedures, withdrawal of consent or any other reason.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-06-25 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- Japan (11):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Gifu, Gifu
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Chuo Ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 11 investigative sites in Japan.
Pre-assignment Details: There was no screening period for this study. At the enrolment visit the patient was consented to the study and eligible participants started their treatment with nilotinib. The parents nilotinib studies are CAMN107G2301 and CAMN107D1201.
Period: Overall Study
Arm/Group | Nilotinib
Started | 15
Completed | 2
Not Completed | 13
Not completed — Disease Progression | 9
Not completed — Adverse Event | 2
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nilotinib
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (13.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of participants with adverse events (AEs) (any AE regardless of seriousness), serious adverse events (SAEs), Fatal SAEs and treatment related AEs.
Time Frame: Adverse events were reported from enrolment until 30 days after last dose of study treatment, up to approximately 10.3 years.
Population: The Safety Set included all participants who received at least one dose of Nilotinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 15
Participants
  Adverse Events | 13
  AEs-Treatment-related | 8
  Serious Adverse Events | 9
  SAEs-Treatment-related | 3
  Fatal SAEs | 1
  Fatal SAEs-Treatment-related | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported from enrolment until 30 days after last dose of study treatment, up to approximately 10.3 years.
Arm/Group | Nilotinib
All-Cause Mortality (participants affected / at risk) | 1/15
Serious Adverse Events (participants affected / at risk) | 9/15
Other Adverse Events (participants affected / at risk) | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=15)
Acute myocardial infarction (Cardiac disorders) | 2
Cataract (Eye disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebellar infarction (Nervous system disorders) | 1
Cerebrovascular insufficiency (Nervous system disorders) | 1
Thrombotic cerebral infarction (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=15)
Anaemia (Blood and lymphatic system disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Cataract (Eye disorders) | 1
Keratitis (Eye disorders) | 1
Polypoidal choroidal vasculopathy (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 2
Enteritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Face oedema (General disorders) | 1
Fatigue (General disorders) | 1
Generalised oedema (General disorders) | 1
Malaise (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Oedema peripheral (General disorders) | 4
Pyrexia (General disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2
Anisakiasis (Infections and infestations) | 1
Influenza (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 5
Pneumonia (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Amylase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Persecutory delusion (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Arterial stenosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/45/NCT01863745/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT01863745/SAP_001.pdf